CLINICAL TRIAL: NCT05296759
Title: A Comparative Study Of Botulinum Toxin Type A Versus Conventional Oral Therapy As A Second Line Treatment Of Diabetic Neuropathy
Brief Title: Botulinum Toxin Type A in Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Eman Hamdy, Principal investigator, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2217
Record Dates: First submitted 2022-03-08; First posted 2022-03-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Botulinum Toxins, Type A; Gabapentin; Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- botulinum toxin A injection (Active Comparator): botulinum toxin A injection
  Interventions: Drug: botulinum toxin A
- gabapentin (Active Comparator): gabapentin
  Interventions: Drug: Gabapentin
- duloxetine (Active Comparator): duloxetine
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: botulinum toxin A — botulinum toxin A injection
  Arms: botulinum toxin A injection
Drug: Gabapentin — Gabapentin oral intake
  Arms: gabapentin
Drug: Duloxetine — Duloxetine oral drug intake
  Arms: duloxetine

SUMMARY:
Background: Diabetes mellitus is commonly complicated by diabetic peripheral neuropathy. Due to common side effects and poor tolerance to medication, poor adherence to medication is common in diabetic peripheral neuropathy. Botulinum toxin A intradermal injection has proved efficacy in cases of diabetic peripheral neuropathy however there is a need to compare its effect with other lines of treatment. The aim of the study was to compare botulinum toxin type a verses conventional oral treatment as a second line treatment of painful diabetic peripheral neuropathy. This study was conducted as a comparative study on 30 patients with type 2 diabetes mellitus proved by nerve conduction study on carbamazepine. Patients were divided randomly into 3 groups. First group was add on duloxetine, second was add on gabapentin and the third group was injected intradermal with botulinum toxin A.

DETAILED DESCRIPTION:
This study is a comparative study on 30 patients with type 2 diabetes mellitus proved by nerve conduction study on carbamazepine. Patients were divided randomly into 3 groups.

First group was add on duloxetine, second was add on gabapentin and the third group was injected intradermal with Botulinum toxin A. Base line Assessment before treatment and follow up assessment as performed The treatment options were explained to the patients and the choice of Botulinum toxin A Intradermal injection was the patient own decision based on inability to be tolerate or adhere to oral treatment.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients type 2 were included on single line of treatment with carbamazepine

Exclusion Criteria:

* any sever medical condition that might interfere with the results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
visual analogue score | 1 week ,4 weeks,12 weeks
  change visual analogue score zero no pain ,10 unbearable pain
Pittsburgh sleep quality index | 1 week ,4 weeks,12 weeks
  change Pittsburgh sleep quality index 0-21 ,above 5 indicates sleep disturbance

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Alexandria university, Alexandria, Egypt